CLINICAL TRIAL: NCT00435188
Title: Life 2: Improving Fitness and Function in Elders
Acronym: Project LIFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: E3386-R
Record Dates: First submitted 2007-02-12; First posted 2007-02-14 (Estimated); Results first posted 2015-01-09 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2015-01

CONDITIONS: Aging; Mobility Limitations
Keywords: Aging; Cost analysis; Counseling; Disabled Persons; Health Promotion; Mobility Limitation; Physical Activity; Primary Care; Randomized Clinical Trial; Veterans
MeSH Terms: conditions — Mobility Limitation; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Behavioral: Multi-component physical activity counseling program A one-year high intensity physical activity counseling program with the following five components: (1) a baseline face-to-face counseling session by the health counselor, (2) follow-up telephone calls by the health counselor biweekly for 6 weekly and then monthly, (3) a one-time physician endorsement of the prescribed exercise regimen in a primary care clinic visit, (4) monthly automated tailored telephone calls from the primary care provider encouraging continued physical activity, and (5) quarterly mailed materials providing personalized feedback
  Interventions: Behavioral: Multi-component physical activity counseling program
- Arm 2 (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Multi-component physical activity counseling program — A one-year high intensity physical activity counseling program with the following five components: (1) a baseline face-to-face counseling session by the health counselor, (2) follow-up telephone calls by the health counselor biweekly for 6 weekly and then monthly, (3) a one-time physician endorsement of the prescribed exercise regimen in a primary care clinic visit, (4) monthly automated tailored telephone calls from the primary care provider encouraging continued physical activity, and (5) quarterly mailed materials providing personalized feedback
  Arms: Arm 1

SUMMARY:
The purpose of this study is to determine whether a 12-month physical activity counseling program, compared to usual care, improves physical performance in a sample of older veterans. The primary physical performance outcome is change in gait speed.

DETAILED DESCRIPTION:
Physical inactivity contributes greatly to the health care burden of older adults and is associated with a high prevalence of functional limitations, morbidity, and disability. Rates of physical inactivity are highest among older adults. Older veterans, compared non-veteran older adults, are more likely to be physically inactive and report more limitations in physical function. Increasing physical activity among older veterans is a promising approach to reduce the burden of chronic disease and its associated functional limitations. The purpose of this study is to determine whether a 12-month physical activity counseling program, compared to usual care, improves physical performance in a sample of older veterans The primary physical performance outcome is change in gait speed. Secondary objectives include examination of the effect of intervention between the two groups (intervention and usual care) on physical activity, self-reported physical function, and health-related quality of life. We also will estimate health care costs between the two groups to determine the short-term economic impact of the counseling in the VHA. Design. Randomized controlled clinical trial. Data collection. All consented patients will receive a baseline computer assisted interview and physical performance test to be repeated quarterly for one-year. The primary outcome is change in gait speed, which is highly predictive of subsequent institutionalization and mortality. Secondary outcome measures include: the SF-36 physical function and other relevant subscales, health-related quality of life, physical activity, self-efficacy, and personal functional goals. Differences between groups for non-routine outpatient clinic use and hospitalization will be explored. The cost of providing an intensive intervention (relative to the cost of usual care) will be calculated relative to functional changes between groups. Individuals randomized to the intervention group will receive a physical activity counseling intervention that includes four components. We will measure and assess change at each endpoint (3,6,9, 12, and 24 months) to determine short and long-term efficacy. Secondary analyses will include: (a) effect of intervention on self-reported physical function, physical activity, personal functional goals, and self-efficacy, and (b) comparison of outpatient clinic use and hospitalization costs between treatment arms relative to intervention costs. Duration Four years. Relevance to the VA. Because approximately 50% of veterans over age 74 have a limiting disability, it is imperative to explore strategies that will alter the course of functional decline of our aging veterans.

ELIGIBILITY:
Inclusion Criteria:

* Age 70 or over
* Followed in VA primary care or geriatrics clinic
* Currently not regularly physically active
* Able to walk 10 meters without human assistance (assistive device acceptable)

Exclusion Criteria:

* Age 70 or over
* Followed in VA primary care or geriatrics clinic
* Currently not regularly physically active
* Able to walk 10 meters without human assistance (assistive device acceptable)
* A terminal diagnosis

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 400 (Actual)
Dates: Start 2004-11; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miriam C. Morey, PhD, Principal Investigator — VA Medical Center
Locations (1):
- VA Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Snyder DC, Morey MC, Sloane R, Stull V, Cohen HJ, Peterson B, Pieper C, Hartman TJ, Miller PE, Mitchell DC, Demark-Wahnefried W. Reach out to ENhancE Wellness in Older Cancer Survivors (RENEW): design, methods and recruitment challenges of a home-based exercise and diet intervention to improve physical function among long-term survivors of breast, prostate, and colorectal cancer. Psychooncology. 2009 Apr;18(4):429-39. doi: 10.1002/pon.1491. PMID 19117329
- [Background] Morey MC, Snyder DC, Sloane R, Cohen HJ, Peterson B, Hartman TJ, Miller P, Mitchell DC, Demark-Wahnefried W. Effects of home-based diet and exercise on functional outcomes among older, overweight long-term cancer survivors: RENEW: a randomized controlled trial. JAMA. 2009 May 13;301(18):1883-91. doi: 10.1001/jama.2009.643. PMID 19436015
- [Result] Morey MC, Peterson MJ, Pieper CF, Sloane R, Crowley GM, Cowper P, McConnell E, Bosworth H, Ekelund C, Pearson M, Howard T. Project LIFE--Learning to Improve Fitness and Function in Elders: methods, design, and baseline characteristics of randomized trial. J Rehabil Res Dev. 2008;45(1):31-42. doi: 10.1682/jrrd.2007.03.0044. PMID 18566924
- [Result] Morey MC, Peterson MJ, Pieper CF, Sloane R, Crowley GM, Cowper PA, McConnell ES, Bosworth HB, Ekelund CC, Pearson MP. The Veterans Learning to Improve Fitness and Function in Elders Study: a randomized trial of primary care-based physical activity counseling for older men. J Am Geriatr Soc. 2009 Jul;57(7):1166-74. doi: 10.1111/j.1532-5415.2009.02301.x. Epub 2009 May 8. PMID 19467149
- [Result] Hall KS, Crowley GM, McConnell ES, Bosworth HB, Sloane R, Ekelund CC, Morey MC. Change in goal ratings as a mediating variable between self-efficacy and physical activity in older men. Ann Behav Med. 2010 Jun;39(3):267-73. doi: 10.1007/s12160-010-9177-5. PMID 20387023
- [Result] Huffman KM, Sloane R, Peterson MJ, Bosworth HB, Ekelund C, Pearson M, Howard T, Pieper CF, Morey MC. The impact of self-reported arthritis and diabetes on response to a home-based physical activity counselling intervention. Scand J Rheumatol. 2010 May;39(3):233-9. doi: 10.3109/03009740903348973. PMID 20429674
- [Result] Huffman KM, Hall KS, Sloane R, Peterson MJ, Bosworth HB, Ekelund C, Pearson M, Howard T, Pieper CF, Morey MC. Is diabetes associated with poorer self-efficacy and motivation for physical activity in older adults with arthritis? Scand J Rheumatol. 2010;39(5):380-6. doi: 10.3109/03009741003605630. PMID 20604671
- [Result] Hall KS, Crowley GM, Bosworth HB, Howard TA, Morey MC. Individual progress toward self-selected goals among older adults enrolled in a physical activity counseling intervention. J Aging Phys Act. 2010 Oct;18(4):439-50. doi: 10.1123/japa.18.4.439. PMID 20956844
- [Result] Hall KS, Sloane R, Pieper CF, Peterson MJ, Crowley GM, Cowper PA, McConnell ES, Bosworth HB, Ekelund CC, Morey MC. Long-term changes in physical activity following a one-year home-based physical activity counseling program in older adults with multiple morbidities. J Aging Res. 2010 Dec 26;2011:308407. doi: 10.4061/2011/308407. PMID 21234104
- [Result] Lum H, Sloane R, Huffman KM, Kraus VB, Thompson DK, Kraus WE, Bain JR, Stevens R, Pieper CF, Taylor GA, Newgard CB, Cohen HJ, Morey MC. Plasma acylcarnitines are associated with physical performance in elderly men. J Gerontol A Biol Sci Med Sci. 2011 May;66(5):548-53. doi: 10.1093/gerona/glr006. Epub 2011 Mar 2. PMID 21367961
- See also: Website containing short physical activity counseling protocols developed for this study. Counseling protocols and physical assessment forms are based on the stage of change transtheoretical models and are modified for older adults. — http://www.research.va.gov/resources/pubs/LIFE-modules.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1, Physical Activity Counseling: Multi-component physical activity counseling program: A one-year high intensity physical activity counseling program with the following five components: (1) a baseline face-to-face counseling session by the health counselor, (2) follow-up telephone calls by the health counselor biweekly for 6 weekly and then monthly, (3) a one-time physician endorsement of the prescribed exercise regimen in a primary care clinic visit, (4) monthly automated tailored telephone calls from the primary care provider encouraging continued physical activity, and (5) quarterly mailed materials providing personalized feedback
- Arm 2, Usual Care: Usual care participants were asked to continue their normal activities and offered a 3-month physical activity counseling program upon completion of the trial
Period: Overall Study
Arm/Group | Arm 1, Physical Activity Counseling | Arm 2, Usual Care
Started | 199 | 199
Completed | 177 | 176
Not Completed | 22 | 23
Not completed — Death | 1 | 6
Not completed — Withdrawal by Subject | 16 | 11
Not completed — Lost to Follow-up | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: Multi-component physical activity counseling program: A one-year high intensity physical activity counseling program with the following five components: (1) a baseline face-to-face counseling session by the health counselor, (2) follow-up telephone calls by the health counselor biweekly for 6 weekly and then monthly, (3) a one-time physician endorsement of the prescribed exercise regimen in a primary care clinic vis
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 199 | 199 | 398
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.7 (5.0) | 77.4 (4.9) | 77.5 (5)
Sex: Female, Male [Count of Participants; unit: Participants] — This study was conducted at a VA Medical Center. Only 3 females were randomized into the study which was not unexpected given the targeted sample and relative paucity of females in VA receiving care in this particular age group at the time. On submitting primary paper, the authors were required to eliminate the females from the study. No females were included in data presented
  Participants
    Female | 0 | 0 | 0
    Male | 199 | 199 | 398
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 48 | 42 | 90
  White | 151 | 157 | 308
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 199 | 199 | 398
Education [Number; unit: participants] — Number of participants completing a categorical level of education as described
  participants
    Less or equal to high school | 91 | 92 | 183
    Some college or trade school | 56 | 52 | 108
    College graduate | 52 | 55 | 107
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 28.9 (4.7) | 29.1 (4.6) | 29 (4.6)
Number of diseases [Mean (Standard Deviation); unit: Diseases] — By self report from a list of 35 conditions adapted from the Older Americans Resources and Services survey
  Diseases | 5.2 (2.5) | 5.5 (2.7) | 5.3 (2.6)
Health quality of life of excellent or very good [Number; unit: participants] — Reported as the number of participants who reported health quality of life as excellent or very good from a 5 point likert scale ranging from poor to excellent
  participants
    Health QOL rated as Excellent or Very Good | 71 | 76 | 147
    Health QOL rated as Good, Fair, or Poor | 128 | 123 | 251
Assistive device [Number; unit: participants] — Number of participants reporting the use of an assistive device
  participants
    Participants reporting assistive device use | 40 | 39 | 79
    Participants reporting no use of assistive devices | 159 | 160 | 319

OUTCOME MEASURES:

1. Primary Outcome: Usual Gait Speed
Description: Best of two trials over 8-foot walk
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 199 | 199
meters/second | 1.03 (0.25) | 1.03 (0.24)

2. Secondary Outcome: Physical Activity Frequency (CHAMPS Questionnaire)
Description: Exercise frequency derived from Community Healthy Activities Model Program for Seniors (CHAMPS) questionnaire; The Champs assesses the frequency of a range of physical activities
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: times per week
Arm/Group | Arm 1, Physical Activity Counseling | Arm 2, Usual Care
Number analyzed (Participants) | 199 | 199
times per week | 15.9 (9.4) | 16.8 (9.8)
Statistical Analysis 1: Comparison: Arm 1, Physical Activity Counseling vs Arm 2, Usual Care; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Omnibus p value for group difference between groups at the end of the study and group by time interaction

3. Secondary Outcome: Physical Activity Frequency (CHAMPS Questionnaire)
Description: as for outcome 2
Time Frame: 3 month
Measure: Mean (Standard Deviation); unit: times per week
Arm/Group | Arm 1, Physical Activity Counseling | Arm 2, Usual Care
Number analyzed (Participants) | 184 | 189
times per week | 22.7 (9.8) | 17.6 (9.4)

4. Primary Outcome: Usual Gait Speed
Time Frame: 3 month
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 184 | 189
meters/second | 1.09 (0.29) | 1.07 (0.28)

5. Primary Outcome: Usual Gait Speed
Time Frame: 12-month
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 178 | 177
meters/second | 1.15 (0.28) | 1.12 (0.25)
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; Omnibus P value reporting overall differences between groups for group and group by time interaction with two degrees of freedom; Test type: Superiority or Other; p = 0.47, Mixed Models Analysis

6. Primary Outcome: Rapid Gait Speed
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 199 | 199
meters/second | 1.56 (0.41) | 1.57 (0.4)

7. Primary Outcome: Rapid Gait Speed
Time Frame: 3-month
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 184 | 189
meters/second | 1.62 (0.5) | 1.58 (0.42)

8. Primary Outcome: Rapid Gait Speed
Time Frame: 12-month
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 178 | 177
meters/second | 1.68 (0.44) | 1.59 (0.42)
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; Omnibus P value for overall difference between groups at the end of the study and group by time interaction on two degrees of freedom; Test type: Superiority or Other; p = 0.04, Mixed Models Analysis

9. Secondary Outcome: Physical Activity Frequency (CHAMPS Questionnaire)
Description: as for outcome 2
Time Frame: 12 month
Measure: Mean (Standard Deviation); unit: times per week
Arm/Group | Arm 1, Physical Activity Counseling | Arm 2, Usual Care
Number analyzed (Participants) | 178 | 177
times per week | 22.4 (12) | 16.8 (9.2)
Statistical Analysis 1: Comparison: Arm 1, Physical Activity Counseling vs Arm 2, Usual Care; Omnibus P value provides the overall differences between groups at the end of the study; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis

10. Secondary Outcome: Self Rated Health
Description: Self-report of overall health, reported as the number of participants reporting health as Excellent or Very good
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 199 | 199
participants
  Overall health is excellent or very good | 71 | 76
  Overall health is good, fair or poor | 128 | 123

11. Secondary Outcome: Self Rated Health
Description: Self-report of overall health, reported as the number of participants reporting health as Excellent or Very good
Time Frame: 3 month
Measure: Number; unit: participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 184 | 189
participants
  Overall health is excellent or very good | 82 | 75
  Overall health is good, fair or poor | 102 | 114

12. Secondary Outcome: Self Rated Health
Description: Self-report of overall health, reported as the number of participants reporting health as Excellent or Very good
Time Frame: 12 month
Measure: Number; unit: participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 178 | 177
participants
  Overall health is excellent or very good | 78 | 70
  Overall health is good, fair or poor | 100 | 107
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; Omnibus P value provides the overall difference between groups at the end of the study; Test type: Superiority or Other; p = 0.29, Mixed Models Analysis

13. Secondary Outcome: Sf-36 Physical Function Subscale
Description: This is a subscale of the SF-36 Medical Outcomes Study. The Physical Function subscale assesses a self-reported ability to perform physical tasks. It is normalized for scores to range from 0 to 100 with a higher score indicating better function.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 199 | 199
units on a scale | 68 (22.2) | 62.9 (23.1)

14. Secondary Outcome: Sf-36 Physical Function Subscale
Description: as for outcome 13
Time Frame: 3 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 184 | 189
units on a scale | 70 (22.4) | 63.1 (24)

15. Secondary Outcome: Sf-36 Physical Function Subscale
Description: as for outcome 13
Time Frame: 12 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 178 | 177
units on a scale | 69.9 (22.1) | 62.7 (23.8)
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; P value provides overall differences between groups at the end of the study; Test type: Superiority or Other; p = 0.35, Mixed Models Analysis

16. Secondary Outcome: 2 Minute Walk
Description: Distance walked in two minutes in meters
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 199 | 199
meters | 146 (36.3) | 145.4 (32.8)

17. Secondary Outcome: 2 Minute Walk
Description: Distance walked in two minutes in meters
Time Frame: 3 month
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 184 | 189
meters | 151.7 (37.8) | 145.6 (34.9)

18. Secondary Outcome: 2 Minute Walk
Description: Distance walked in two minutes in meters
Time Frame: 12 month
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 178 | 177
meters | 150.9 (38.5) | 147.5 (34.7)
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; P value provides the overall differences between groups at the end of the study; Test type: Superiority or Other; p = 0.08, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Arm 1, Physical Activity Counseling | Arm 2, Usual Care
Serious Adverse Events (participants affected / at risk) | 0/199 | 0/199
Other Adverse Events (participants affected / at risk) | 3/199 | 0/199
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1, Physical Activity Counseling (N=199) | Arm 2, Usual Care (N=199)
minor injury (Musculoskeletal and connective tissue disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No